CLINICAL TRIAL: NCT05438459
Title: Clinical Trial of Repeated Intraperitoneal Administration of GAIA-102 in Patients With Advanced Gastrointestinal Cancer (Gastric Cancer / Pancreatic Cancer) of Microsatellite Stable (MSS) With Malignant Ascites (Phase I / II Investigator-initiated Clinical Trial) (GAIA-102-PD Clinical Trial)
Brief Title: GAIA-102 Intraperitoneal Administration in Patients With Advanced Gastrointestinal Cancer of Microsatellite Stable With Malignant Ascites
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kyushu University (Other)
Collaborators: GAIA BioMedicine Inc. (Industry); Toho University - Omori Medical Center (Unknown); Jichi Medical University (Other); Kindai University Hospital (Unknown); Teikyo University Hospital (Unknown); Kansai Medical University Hospital (Unknown); Kyushu Cancer Center (Unknown)
Responsible Party: Principal Investigator, EijiOki, Lecturer, Kyushu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTR024-001
Record Dates: First submitted 2022-06-13; First posted 2022-06-30 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Gastric Cancer; Pancreatic Cancer
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GAIA-102 as a monotherapy (Experimental): GAIA-102: 1 vial (2 x 10^8 cells) as dose at a fixed dose, on 1 to 3 times by weekly for 3 consecutive weeks.
  Interventions: Biological: Phase I part; Biological: Phase II part
- GAIA-102 and pembrolizumab in combination (Experimental): GAIA-102: 1 vial (2 x 10^8 cells) as dose at a fixed dose, on 1 to 3 times by weekly for 3 consecutive weeks.
  Pembrolizumab：200 mg on Day 1.
  Interventions: Biological: Phase I part; Biological: Phase II part
- Ttrifluridine/tipiracil hydrochloride (FTD/TPI) as the standard therapy group (Experimental): Trifluridine/tipiracil hydrochloride (FTD/TPI) : Trifluridine/tipiracil hydrochloride (FTD/TPI) will be administered orally twice daily for 5 consecutive days, followed by a 2-day rest period. This cycle will be repeated twice, followed by a 14-day rest period. One course consists of this schedule, and the treatment will be repeated in cycles.
  Interventions: Biological: Phase II part

INTERVENTIONS:
Biological: Phase I part — Administration of GAIA-102 as a monotherapy or GAIA-102 and pembrolizumab in combination.
  Arms: GAIA-102 and pembrolizumab in combination; GAIA-102 as a monotherapy
Biological: Phase II part — Patients will be randomly assigned to receive either GAIA-102 monotherapy or GAIA-102 in combination with pembrolizumab at the recommended dosing regimen confirmed in the Phase I part, or to receive standard therapy.
  For patients with gastric cancer, the standard therapy group will receive trifluridine/tipiracil hydrochloride (FTD/TPI) only.

SUMMARY:
Phase I Part :

Confirm the safety of GAIA-102 as a monotherapy or GAIA-102 and pembrolizumab in combination for advanced gastrointestinal cancer of microsatellite stable with malignant ascites, and determine the recommended number of doses for Phase II part.

Phase II Part :

Research the efficacy and safety of as a monotherapy or GAIA-102 and pembrolizumab for advanced gastrointestinal cancer of microsatellite stable with malignant ascites at the recommended dose of GAIA-102 decided in the Phase I part.

ELIGIBILITY:
Inclusion Criteria:

1. Unresectable or advanced recurrent gastric cancer with evident peritoneal dissemination on imaging, or with ascites, as well as unresectable or advanced recurrent pancreatic cancer.
2. Phase I:

   Patients with gastric cancer who have received 3 or more prior chemotherapy regimens and are refractory or intolerant to these therapies, and patients with pancreatic cancer who have received 2 or more prior chemotherapy regimens and are refractory or intolerant to these therapies.

   Phase II:

   Patients with gastric cancer who have received 2 or more prior chemotherapy regimens, including at least 1 regimen containing an immune checkpoint inhibitor, and are refractory or intolerant to these therapies, and patients with pancreatic cancer who have received 1 or more prior chemotherapy regimens and are refractory or intolerant to these therapies.
3. Abdominal port placement is possible
4. No medical history of serious side effects or allergic reactions to pembrolizumab (only for patients in the pembrolizumab combination cohort)
5. Diagnosed gastric adenocarcinoma or pancreatic cancer with by histological or cytological examination
6. The patient has been confirmed to be "negative (not MSS = MSI-high)" by microsatellite instability (MSI) testing, or "proficient mismatch repair (pMMR)" by mismatch repair protein immunohistochemistry testing
7. The Eastern Cooperative Oncology Group (ECOG) performance status(PS) at the time of informed consent meets the following conditions.

   * Phase I ：0-2
   * Phase II ：0-1
8. Patient aged 20years or older
9. Adequate major organs (bone marrow, heart, lungs, liver, kidneys, etc.) function:

   * Neutrophil ≧1,500/mm3
   * hemoglobin ≧8.0 g/dL
   * Platelet ≧75,000/mm3
   * PT-INR≦ 1.5
   * AST, ALT≦ 3 times the upper limit of reference value
   * T-Bil≦ 2 times the upper limit of reference value (T-Bil ≦ 3.0mg/dL , when drainage for obstructive jaundice)
   * eGFR ≧30mL/min/1.73m2
10. Expected to survive for 3 months or more at the enrollment
11. Written informed consent

Exclusion Criteria:

1. Untreated cranial metastases.
2. Diagnosed with meningeal carcinomatosis
3. Received allogeneic hematopoietic stem cell transplantation
4. Participated in other clinical trials / clinical trials within 30 days prior to obtaining written consent and used or had used the investigational product or investigational equipment.
5. Existence or suspected active autoimmune disease
6. Continued systemic immunosuppressive therapy with corticosteroids in excess of 10 mg / day in terms of prednisolone or other immunosuppressants within 14 days prior to investigational product administration
7. Symptomatic interstitial pneumonia, or even if it is not symptomatic, it may interfere with diagnostic imaging in detecting new pneumonitis caused by the investigational product used in the clinical trial.
8. Have active double cancer and need treatment for the double cancer
9. Requires treatment as shown in "Unacceptable Combination / Supportive Therapy" during the clinical trial period
10. Have a medical history of severe hypersensitivity to immune checkpoint inhibitors or immune-related adverse events requiring treatment
11. Have one of the following complications

    * Complication of cerebrovascular disorder with symptoms or history within 6 months before the enrollment
    * Active gastrointestinal perforation, fistula, diverticulitis
    * Symptomatic congestive heart failure
    * Bleeding tendency
    * Presence of blood clots that may cause embolism on the image
    * Unhealed fractures (excluding compression fractures associated with osteoporosis) or severe wounds requiring medical treatment
    * Uncontrollable digestive ulcer
    * Active infectious diseases requiring intravenous administration of antibiotics, antifungal agents or antiviral agents
    * HIV antibody positive
12. At the time of the enrollment, the period from the following prior treatment or the end of treatment has not passed.

    * Surgery (including exploratory laparotomy / examination laparoscope): 2 weeks
    * Palliative radiotherapy: 1 week
    * Thoracic drainage: 1 week
    * Pretreatment antineoplastic (from the last administration): 3 weeks
    * Biopsy with incision, thoracic biopsy, treatment for trauma (excluding patients without wound healing), etc : 2 weeks
13. Scheduled thoracotomy or abdominal surgery during the clinical trial period
14. It is judged that it is difficult to enroll in this study due to clinically significant mental illness.
15. Pregnant women, lactating women, women who are currently pregnant, or have no intention of contraception for 4 months after consent is obtained.
16. Allergic to antibiotics and foreign animal-derived ingredients (pig and mouse)
17. Difficult to participate in the trial by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants of Dose Limiting Toxicity (DLT) with GAIA-102 (Phase I) | Cycle 1 (Cycle period is 28 days)
  DLT was evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 and is defided following events: 1. Grade 4 hemotoxicity or hemotoxicity requiring blood transfusion. 2. Grade 3 or higher non-hematoxicity
Frequency and severity of adverse events(Phase I) | 2 year
Overall survival period in patients with gastric cancer (Phase II) | up to 4 years
One-year survival rate in patients with pancreatic cancer (PhaseⅡ) | 1 year

SECONDARY OUTCOMES:
Objective Response Rate （ORR) and Disease Control Rate (DCR)(Phase I) | Week 24
Progression-free Survival(Phase I) | 2 year
Overall Survival Period(Phase I) | 2 year
Pharmacokinetics of GAIA-102(Phase I) | pre-dose
  The following metrics were meassured as pharmcokinetics; Cmax: The peak plasma concentration of a drug after administration.; tmax. : Time to reach Cmax; Cmin: The lowest (trough) concentration that a drug reaches before the next dose is administered.
Biomarker of GAIA-102(Phase I) | pre-dose
  Protein expression levels are measured in ascites and blood as biomarkers. The following are the markers to be measured; CCL3/CCL4/CCL5/CCL20/CXCL9/CXCL10/CXCL11
Objective Response Rate Disease Control Rate(Phase II) | up to 4 years
Progression-free Survival (Phase II) | up to 4 years
Objective Response Period and Period until Objective Response (Phase II) | up to 4 years
One-year survival rate in patients with gastric cancer (Phase II) | 1 year
Overall survival period in patients with pancreatic cancer (Phase II) | up to 4 years
Frequency and severity of adverse events (Phase II) | up to 4 years
Biomarker of GAIA-102(Phase II) | pre-dose
  Protein expression levels are measured in ascites and blood as biomarkers. The following are the markers to be measured; CCL3/CCL4/CCL5/CCL20/CXCL9/CXCL10/CXCL11

CONTACTS AND LOCATIONS:
Locations (1):
- Kyushu University Hospital, Fukuoka, Fukuoka, Japan